CLINICAL TRIAL: NCT03494439
Title: Prevalence of Anterior Open Bite in a Group of Egyptian Children Aged Eight Years and Above: A Cross Sectional Study
Brief Title: Prevalence of Anterior Open Bite in a Group of Egyptian Children Aged Eight Years and Above
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant Mohamed Elmesbahy, B.D.S 2013, Cairo University
Other Study IDs: CEBD-CU-2018-04-02
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Anterior Open Bite

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the prevalence of anterior open bite and its etiological factors in a group of Egyptian children aged 8 years and above. patients who met the eligibility criteria will be given a questionnaire to fill followed by obtaining casts stabilized into occlusion to obtain the vertical and horizontal relationships.

ELIGIBILITY:
Inclusion Criteria:

* Medically free children aged 8 years and above, both genders and cooperative parents and children

Exclusion Criteria:

* Presence of orthodontic appliance and parents refuse to participate

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptian children aged 8 years and above, from the Out Patients' clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Anterior Open bite | 1 year
  Overbite and Overjet measurement by obtaining a cast to determine anterior open bite in millimeters

SECONDARY OUTCOMES:
Its different etiological factors | 1 year
  Asking patient/ caregiver through a (Questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided